CLINICAL TRIAL: NCT03282929
Title: An Single-dose, Open Label, Randomized Cross-over Study to Explore the Pharmacokinetics and Pharmacodynamics of Epinephrine in Healthy Male and Female Subjects With Different Skin to Muscle Depth (STMD)
Brief Title: Study to Explore the Pharmacokinetics and Pharmacodynamics of Epinephrine in Healthy Male and Female Subjects With Different Skin to Muscle Depth (STMD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N-A-PH1-15-050
Record Dates: First submitted 2017-07-21; First posted 2017-09-14 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Anaphylaxis
MeSH Terms: conditions — Anaphylaxis

STUDY DESIGN:
Intervention Model Description: Pharmacokinetics and pharmacodynamics of epinephrine in healthy male and female subjects with different skin-to-muscle depth (STMD) of the thigh after injections with four different marketed auto-injectors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Part 1 Group 1 (Experimental): A single dose of 500 μg epinephrine (0.5 mL Suprarenin®) will be administered i.m. and s.c. by using a needle and a syringe in randomized order.
  Interventions: Device: Part 1
- Part 2 group 1 (Experimental): 300 μg epinephrine auto-injector (Emerade, Bausch and Lomb, 23 mm needle length)
  Interventions: Device: Part 2 Group 1
- Part 2 Group 2 (Experimental): 500 μg epinephrine auto-injector (Emerade, Bausch and Lomb, 23 mm needle length)
  Interventions: Drug: Part 2 group 2
- Part 2 Group 3 (Experimental): 300 μg epinephrine auto-injector (Fastjekt, MEDA Pharma, 16 mm needle length)
  Interventions: Device: Part 2 group 3
- Part 2 Group 4 (Experimental): 300 μg epinephrine auto-injector (Jext, Alk-Abelló, 15 mm needle length)
  Interventions: Device: Part 2 Group 4

INTERVENTIONS:
Device: Part 1 — A single dose of 500 μg epinephrine (0.5 mL Suprarenin®) will be administered i.m. and s.c. by using a needle and a syringe in randomized order
  Other Names: Group 1
  Arms: Part 1 Group 1
Device: Part 2 Group 1 — 300 μg epinephrine auto-injector (Emerade, Bausch and Lomb, 23 mm needle length)
  Other Names: Group 1
  Arms: Part 2 group 1
Drug: Part 2 group 2 — 500 μg epinephrine auto-injector (Emerade, Bausch and Lomb, 23 mm needle length)
  Other Names: Group 2
  Arms: Part 2 Group 2
Device: Part 2 group 3 — 300 μg epinephrine auto-injector (Fastjekt, MEDA Pharma, 16 mm needle length)
  Other Names: Group 3
  Arms: Part 2 Group 3
Device: Part 2 Group 4 — 300 μg epinephrine auto-injector (Jext, Alk-Abelló, 15 mm needle length)
  Other Names: Group 4
  Arms: Part 2 Group 4

SUMMARY:
A single dose, open label, randomized cross-over study to explore the pharmacokinetics and pharmacodynamics of epinephrine in healthy male and female subjects

DETAILED DESCRIPTION:
A single dose, open label, randomized cross-over study to explore the pharmacokinetics and pharmacodynamics of epinephrine in healthy male and female subjects with different skin-to-muscle depth (STMD) of the thigh after injections with four different marketed auto-injectors

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, between 18 and 54 years of age (inclusive).
2. Subjects who are able and willing to give written informed consent.
3. Body mass index (BMI) between 28.0 and 40.0 kg/m² (inclusive). Weight on Day -1 may not have changed by more than 3 kg compared to screening.
4. Compressed STMD of 10 mm and above (Part 1+2).
5. Non-smoker for at least 6 months.

Exclusion Criteria:

1. Receipt of medication (prescription or non-prescription) within 14 days prior to the planned drug administration, except for occasional use of paracetamol or ibuprofen.
2. Receipt of any of the following medications within the previous 6 months; beta adrenergic blockers, tricyclic antidepressants, monoamine oxidase inhibitors and catechol-O-methyl transferase inhibitors, methylphenidate, amphetamines, any drugs that may sensitize the heart to arrhythmias, including digitalis and quinidine.
3. History or current evidence of a clinically significant disease including, but not limited to: cardiovascular, hepatic, renal, hematological, neuropsychological, endocrine, gastrointestinal or pulmonary diseases especially asthma bronchiale. Significant is defined as any disease that, in the opinion of the investigator, would put the safety of the subject at risk through participation, or which could affect the endpoint analysis if the disease/condition exacerbated during the study.

   History or presence of silent infections, including positive tests for HIV1, HIV2, Hepatitis B or C.
4. Presence of any disease or condition known to interfere with the absorption, distribution, metabolism or excretion of drugs.
5. Hypersensitivity to epinephrine or any of the excipients (e.g. metabisulphite).

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2018-09-28 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Cmax | 14 days
  Maximum observed drug concentration
tmax | 14 days
  Time of the maximum drug concentration (obtained without interpolation). If the maximum value occurs at more than one time point, tmax is defined as the first time point with this value.

CONTACTS AND LOCATIONS:
Overall Officials: Beate Klaus, MD, Principal Investigator — Baush and Lomb
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Wegenerstrasse 13, Germany